CLINICAL TRIAL: NCT05779592
Title: An Observational Study Evaluating Treatment Situations of Adjuvant Nivolumab for Muscle-invasive Urothelial Carcinoma in Japan
Brief Title: A Study to Evaluate Nivolumab in Japanese Participants With Muscle-invasive Urothelial Carcinoma
Acronym: ANNIVERSARY
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6H7
Record Dates: First submitted 2023-02-24; First posted 2023-03-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Muscle-invasive Urothelial Carcinoma
Keywords: UC; Nivolumab; UTUC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Cohort 1: Muscle-invasive Urothelial Carcinoma Participants who received nivolumab as adjuvant treatment at least once from March 28, 2022 to December 31, 2023

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and actual treatment status of nivolumab administered as an adjuvant treatment for participants with muscle-invasive urothelial carcinoma (MIUC), including bladder, renal pelvis, and ureteral cancer, in a Japanese real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically definitive diagnosis of MIUC at each study site and who must have received nivolumab after radical resection
* Must present at least once to the study site after nivolumab treatment or must have survival data

Exclusion Criteria:

* Participants who underwent only partial resection for MIUC
* Participants treated with chemotherapy, radiotherapy, biologics (anticancer agents), intravesical chemotherapy, or Bacillus Calmette-Guérin therapy from the time of radical resection of MIUC to the start of nivolumab
* Participants previously treated with immune checkpoint inhibitors prior to nivolumab treatment

Other protocol-specific inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received adjuvant treatment with nivolumab for Muscle-invasive Urothelial Carcinoma (MIUC) at least once from March 28, 2022 to December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 4 years
  The time from the date of nivolumab initiation to the date of first recurrence (urothelial local recurrence, non-urothelial local recurrence, or distant recurrence) or death from any cause as an event, whichever occurs first.
Non-urothelial tract recurrence free survival (NUTRFS) | Up to 4 years
  The time from the date of nivolumab initiation to the date of first recurrence (local or distant non-urothelial recurrence) or death from any cause as an event, whichever occurs first.
Number of participants with adverse events (AEs) | Up to 4 years
Number of participants with treatment-related adverse events (TRAEs) | Up to 4 years
Actual treatment status: dosing frequency | Up to 4 years
Actual treatment status: treatment duration | Up to 4 years
  The time from the start date of nivolumab administration to the last administration date
Actual treatment status: treatment completion rate | Up to 4 years
  The treatment completion rate will be calculated* according to the following formula:
  Treatment completion rate (%)=(Patients who completed treatment)/(All eligible patients)×100
Actual treatment status: reason for discontinuation | Up to 4 years

SECONDARY OUTCOMES:
DFS | Up to 4 years
  The time from the date of nivolumab initiation to the date of first recurrence (urothelial local recurrence, non-urothelial local recurrence, or distant recurrence) or death from any cause as an event, whichever occurs first.
NUTRFS | Up to 4 years
  The time from the date of nivolumab initiation to the date of first recurrence (local or distant non-urothelial recurrence) or death from any cause as an event, whichever occurs first.
Number of participants with AEs | Up to 4 years
Number of participants with TRAEs | Up to 4 years
Actual treatment status: dosing frequency | Up to 4 years
Actual treatment status: treatment duration | Up to 4 years
  The time from the start date of nivolumab administration to the last administration date
Actual treatment status: treatment completion rate | Up to 4 years
  The treatment completion rate will be calculated* according to the following formula:
  Treatment completion rate (%)=(Patients who completed treatment)/(All eligible patients)×100
Actual treatment status: reason for discontinuation | Up to 4 years
Overall survival (OS) | Up to 4 years
  The time from the date of nivolumab initiation to the date of death from any cause
Disease-specific survival (DSS） | Up to 4 years
  The time from the date of nivolumab initiation to the date of death due to the primary disease
Number of participants with immune-mediated adverse events (IMAEs) according to the Common Terminology Criteria for Adverse Events (CTCAEs) version 5.0 | Up to 4 years
Number of participants with TRAEs leading to treatment discontinuation | Up to 4 years
Actual treatment status: treatment continuation rate | Up to 4 years
  Treatment continuation rate (%)=(Patients continuing treatment at the timepoint)/(All eligible patients)×100
Actual treatment status: dosing intensity | Up to 4 years
  Dose intensity (%)=(Actual dose)/(Total dose planned)×100
Post-recurrence treatment status: The number of participants transitioning to treatment | Up to 4 years
  The proportion of eligible patients who completed and started treatment after recurrence.
The number of participants with complete response (CR) due to treatment relative to those with evaluable disease who were treated after recurrence | Up to 4 years
The number of participants with partial response (PR) due to treatment relative to those with evaluable disease who were treated after recurrence | Up to 4 years
The proportion of participants with complete response (CR) due to treatment relative to those with evaluable disease who were treated after recurrence | Up to 4 years
The proportion of participants with partial response (PR) due to treatment relative to those with evaluable disease who were treated after recurrence | Up to 4 years
The number of participants in each BOR category (CR/PR/stable disease (SD)/progressive disease (PD)/ not evaluated (NE)) receiving treatment after recurrence | Up to 4 years
The proportion of eligible participants with evaluable disease | Up to 4 years
Duration of treatment | Up to 4 years
  The time from the start date of treatment administration to the last administration date after recurrence.
Time to treatment | Up to 4 years
  The time from the start date of nivolumab to the start date of treatment after recurrence.
Estimated glomerular filtration rate (eGFR) | Up to 4 years
  Measured before NAC, before radical resection, immediately before nivolumab treatment, at the time of recurrence, or at the start of post-recurrence treatment
The regimen of Neoadjuvant chemotherapy (NAC) performed prior to radical resection in eligible participants | Up to 4 years
The number of cycles of Neoadjuvant chemotherapy (NAC) performed prior to radical resection in eligible participants | Up to 4 years
The clinical stage prior to NAC | Up to 4 years
The pathologic stage at the time of radical resection | Up to 4 years
Treatment completion rate (%) | Up to 4 years
  (Participants who completed treatment)/(All eligible participants)x100

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, City, State, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm